CLINICAL TRIAL: NCT03867422
Title: Changes in Brain Tissue Pulsatility With Musical Stimuli
Acronym: M-PULSE
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI19-M-PULSE
Record Dates: First submitted 2019-03-04; First posted 2019-03-08 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Music Perception is well known to elicit emotions and neuronal activations. Changes in the cerebrovascular physiology have also been found in emotional tasks but only few studies have investigated markers of cerebrovascular physiology in a music task and no study has used the Ultrasound method of Tissue Pulsatility Imaging (TPI) in a music task. The use of TPI to measure reactivity of Brain Tissue Pulsatility Imaging (BTP) could further elucidate the cerebral basis of music perception.

ELIGIBILITY:
Inclusion Criteria:

* more or equal 18 years-old and less or equal 45 years-old
* no known hearing problem

Exclusion Criteria:

* professional musician
* history of neurologic, psychiatric or cadiologic disease
* treatment which could impact parameters of brain tissue pulsatility and peripheral nervous system
* opposition to use the data

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
amplitude of variations in brain tissue pulsatility | Baseline
  in micrometers

SECONDARY OUTCOMES:
heart rate | Baseline
  beat by minute
breathing rate | Baseline
  Frequency
skin conductance | Baseline
  in milliVolt
score of barcelona music reward questionnary (BMQR) | Baseline
  BMQR: Barcellona Music Reward Questionnaire for the evaluation of musical anhedonia;
  * Only the total score of musical reward will be reported; for total score, minimum value is 20, maximum value is 100. Values under 40 represent low values in the overall score; values above 60 indicate high values in the overall score;
  * High global score (>60) represents a better outcome; low global score (<40) represents a worse outcome, notably an impairment in music reward processing;
  * The overall score is computed by adding raw scores of the items (except for items 2 and 5, which need to be reversed).

CONTACTS AND LOCATIONS:
Locations (1):
- DESMIDT, Tours, France

IPD SHARING:
Plan to Share IPD: No